CLINICAL TRIAL: NCT06461611
Title: Effect of Health Diary on Self-management in Adolescent Patients With Orthodontic Fixed Appliance: A Randomized Controlled Trial
Brief Title: Effect of Health Diary on Self-management in Adolescent Patients With Fixed Orthodontic Appliance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Association Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CJ-KQEC-2024-48-01
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Oral Hygiene; Self-Management
Keywords: Malocclusion; Fixed Orthodontic Treatment; Adolescent; Self-Management; Self-Efficacy; Health Diary; Oral Health-Related Quality of Life; Oral Hygiene
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Investigator
Masking Description: A qualified examiner blinded to individual subject treatment assignments performed the oral hygiene status index （SBI and PLI）on subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients in the control group will receive traditional health education, which consist of routine oral health education and oral health instructions during their visits for orthodontic treatment.
  Interventions: Behavioral: Traditional Health Education
- Intervention Group (Experimental): Patients in the intervention group will receive a health diary to plan and clock for their fixed orthodontic self-management behaviors in addition to the traditional health education.
  Interventions: Behavioral: Health Diary Program

INTERVENTIONS:
Behavioral: Health Diary Program — The health diary is constructed based on the theory of health action process approach, which is used to plan and clock for self-management behaviors of adolescent patients during fixed orthodontic treatment.
  Arms: Intervention Group
Behavioral: Traditional Health Education — Traditional health education is that the nurse orally teaches the patient about fixed orthodontic knowledge, and the patient obtains a paper information.
  Arms: Control Group

SUMMARY:
This study aims to use two-arm randomized clinical trials to evaluate the effectiveness of the health diary in helping adolescents wearing fixed orthodontic appliances improve their oral hygiene status, self-management skills, oral health-related quality of life, self-efficacy, intention，number of breakages, and on-time and return visit status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malocclusion eligible for fixed appliance orthodontic treatment;
* The age of patients ranged from 12 to 18 years;
* The patients received orthodontic treatment for the first time;
* The patient was alert and had no cognitive or psychiatric impairment;
* The patient was able to read and fill out the questionnaires, and had good listening, speaking and understanding skills in Chinese.

Exclusion Criteria:

* The patient's disease was diagnosed as jaw deformity associated with other diseases. Malocclusion secondary to trauma, tumor, cleft lip and palate;
* Patients treated with orthodontic-orthognathic surgery;
* The patient currently participating in other oral related intervention studies.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | Change from baseline plaque index at 24-weeks follow-up.
  Ramfjord index teeth (16, 21, 24/25, 36, 41, 44/45) were selected. After staining with plaque stain, the plaque area of mesial, middle buccal, distal buccal and lingual surface of each tooth was examined, and the average value of the four dental surfaces was recorded. Finally, the PLI score was calculated by adding the index teeth and dividing by the number of teeth examined.
Bleeding Index | Change from baseline plaque index at 24-weeks follow-up.
  It is a combination of visual examination and probing. The probe was inserted into the gingival sulcus for 1 second and then removed. After 30 seconds, the gingival bleeding and the degree of bleeding were observed. Ramfjord index teeth were selected, namely 16, 21, 24/25, 41, 44/45.The detection sites of each index tooth included 6 sites in the mesial, distal and central of the buccal and lingual surface. The sum of the scores of the examined teeth and then divided by the number of examined teeth were used to determine the SBI score of the patient.

SECONDARY OUTCOMES:
Self-Management Ability | Change from baseline plaque index at 24-weeks follow-up.
  The self-management Ability scale for Adolescent Patients with fixed orthodontics was used for evaluation. The higher the score of the scale, the higher the self-management ability.
Self Efficacy | Change from baseline plaque index at 24-weeks follow-up.
  Self-efficacy in this study refers to oral health care self-efficacy, as assessed by the Oral Health Care Self-efficacy Scale (SEOH-C), with higher scale scores indicating greater self-efficacy.
Oral Health Related Quality of Life | Change from baseline plaque index at 24-weeks follow-up.
  OHRQoL was assessed using the Oral Health Impact Profile 14 (OHIP-14), with higher score indicating lower oral health-related quality of life.
The number of appliance damage in each follow-up period | The number of appliance damage in each follow-up period change over 24 weeks during intervention from baseline.
  The compliance of diet management was indirectly evaluated by monitoring the number of appliance damage. The number of appliance damage between the date of the current visit and the expected date of the next visit was recorded as follows: number of appliance damage = number of brackets lost + number of buccal canals lost + number of archwires broken + number of archwires slipped out of the bracket.
On-time follow-up visits | On-time follow-up visits change over 24 weeks during intervention from baseline.
  In this study, on-time follow-up was defined as the patients attending the follow-up date according to the doctor's advice, and the treatment content on the day of the follow-up visit was adjustment of appliance force, etc. The following orthodontic emergencies were excluded: the treatment only involved the patients who did not meet the doctor's advice for the follow-up due to pain and discomfort caused by bracket loss, buccal canal loss, arch wire fracture, or arch wire slipping out of the bracket groove, and the routine orthodontic follow-up was not involved during the treatment. The on-time return visit was judged according to the interval days between the date of the patient's doctor's advice and the actual date of return visit, and the absolute value of the date of the doctor's advice minus the actual date of return visit was recorded. A difference of "0" was marked as "very punctual"; 0 to 14 was scored as "on time" and more than 14 as "not on time".

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No